CLINICAL TRIAL: NCT05463432
Title: An Open-label Phase 1a Study of the Safety and Tolerability of HR19024 Injection in Subjects With Advanced Solid Tumor
Brief Title: A Study of HR19024 in Subjects With Advanced Solid Tumor
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Hengrui Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HR19024-101
Record Dates: First submitted 2022-07-07; First posted 2022-07-19 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Advanced Solid Tumor

STUDY DESIGN:
Intervention Model Description: HR19024 for all enrolled subjects
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HR19024 (Experimental): Part 1: Dose escalation of HR19024 montherapy for advanced solid tumor Part 2：PK expansion of HR19024 montherapy for advanced solid tumor Part 3: Efficacy expansion of HR19024 montherapy for advanced solid tumor
  Interventions: Drug: HR19024

INTERVENTIONS:
Drug: HR19024 — Intravenous infusion

SUMMARY:
To evaluate the safety，tolerability，pharmacokinetic characteristics and preliminary efficacy of HR19024 injection in the treatment of advanced solid tumor

ELIGIBILITY:
Inclusion Criteria:

1. ECOG performance status 0 or 1
2. Histologically confirmed advanced solid tumor
3. Life expectancy of greater than or equal to (>=) 12 weeks
4. At least one measurable lesion is present according to the efficacy evaluation criteria for solid tumors (RECIST 1.1)
5. Able and willing to provide a written informed consent

Exclusion Criteria:

1. Subjects with unresolved toxicity （> CTCAE G1）of prior therapy at the time of enrolment
2. Subjects who had received anti-tumor treatments such as surgery, chemotherapy, radiotherapy recently

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2022-08-10 (Actual); Primary Completion 2024-10-22 (Actual); Study Completion 2024-10-22 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) of HR19024 | 21-day cycle (tri-weekly)

SECONDARY OUTCOMES:
Response rate (RR) | up to 6 months following the date the last patient was randomized
Disease Control Rate | up to 6 months following the date the last patient was randomized
Duration of Response | up to 6 months following the date the last patient was randomized
Progression free survival (PFS) | up to 6 months following the date the last patient was randomized

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided